CLINICAL TRIAL: NCT07161024
Title: AR Projections for Eye-gaze Evaluation in Phantoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Vanderbilt University (Other); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Nicholas Kavoussi, Assistant Professor Department of Urology, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 231997; 1R21EB035783-01 (NIH)
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Kidney Stones
Keywords: Kidney Stones; Augmented Reality; Gaze Guidance
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AR Marker Test (Experimental): Each user performs a kidney stone identification task in phantoms with each of three augmented reality markers, and without any marker. The phantoms and markers ordering are randomized to reduce learning effect.
  Interventions: Device: Augmented reality

INTERVENTIONS:
Device: Augmented reality — Augmented reality markers of different designs are tested to evaluate how they affect trainee performance.

SUMMARY:
This project aims to develop an augmented reality (AR) tool to enhance skill acquisition for endoscopic kidney stone surgery. Of the 100,000 patients who undergo an endoscopic kidney stone treatment annually in the United States, 25% will require a repeat stone surgery within 20 months of their index surgery. The repeat stone surgery rate is almost completely driven by postoperative residual stone fragments, which lead to ureteral obstruction, causing pain, urinary tract infection, and kidney injury. One significant factor that contributes to residual stone fragments is limited visualization of the entire collecting system - a skill directly associated with surgeon experience. This leads to novice surgeons having a much higher recurrence rate than experienced ones. As the incidence of kidney stone disease continues to increase (prevalence of 10%, incidence of 1116 per 100,000), improved endoscopic surgical training is required to improve outcomes of stone surgeries and minimize complications by improving stone-free rate.

Currently, skill assessment during endoscopic stone surgery is limited. There are no objective metrics for endoscopic surgery to assess skill. The only feedback trainees get is in the form of verbal communication from expert surgeons, usually after the conclusion of surgery. Thus, most feedback is synoptic and limited in facilitating skill acquisition. Operative time and patient safety concerns restrict the amount of active, real-time feedback given during a case for skill acquisition. Endoscopic kidney stone surgery is uniquely challenging given the small depth and field of view of current endoscopes, which complicate the complete visualization of the entire collecting system.

Navigation of the collecting system relies on mentally mapping preoperative imaging to the endoscopic surgical field. Success in mapping relies on hand-eye coordination, memory, and spatial reasoning, which are gained through practice. Thus, there is a need for tools that facilitate endoscopic surgical skill acquisition.

The overarching hypothesis for this research is that surgical skill acquisition and outcomes for endoscopic kidney stone surgery can be improved by analyzing eye gaze data and using expert gaze to guide surgical trainees intraoperatively. Eye gaze guidance has been shown to lead to better skill acquisition in virtual reality surgical tasks compared with motion guidance alone. The proposed system would provide real-time education for trainees during endoscopic stone surgery, such as through head-mounted displays (i.e., the Microsoft HoloLens 2). The investigators have previously demonstrated eye gaze sharing in phantoms. By implementing this system in the operating room (OR), the investigators would be able to instill durable skill acquisition in trainees. The investigators will also implement the NASA-task load index for the trainees to gauge the usability of the system.

DETAILED DESCRIPTION:
Specifically for this study, the investigators are asking each participant, all surgical trainees, to explore four phantom kidneys with stones added and count the number of stones. For each kidney phantom, the participants will have either one of three augmented reality markers to show where an expert is looking, or they will not have any visual guidance (standard of care). In all cases, the participants get verbal feedback from the expert surgeon. The goal is to compare the effect of the design of the AR marker on the trainee's performance in exploring the kidney phantom.

ELIGIBILITY:
Inclusion Criteria:

* Urology residents at Vanderbilt University Medical Center

Exclusion Criteria:

-

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
NASA Task Load Index | 1 m in
  Conducted after each trial for subjective feedback

SECONDARY OUTCOMES:
Kidney exploration | 1-10 min
  Percentage of kidney that was visualized
Stone count | 1-10 min
  Number of stones seen
Gaze metrics | 1-10 min
  Extracted from eye-camera recording from the HoloLens 2
Completion time | 1-10 min
  Time for the stone identification task

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share the endoscope video and eye-gaze information from the study, and associated metadata, including the study protocol.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The manuscript describing the study method and findings has been accepted for publication and will appear in September. We plan to upload the data to the NIDDK repository by December 2025. We foresee both being available indefinitely.
Access Criteria: Anyone can access the research manuscript with aggregate results. Access to individual data will be controlled through the NIDDK repository and available only for research purposes.

DOCUMENTS (1):
  • Informed Consent Form (2025-05-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT07161024/ICF_001.pdf